CLINICAL TRIAL: NCT05780060
Title: Multiple Organized Systems for Engaging Stroke (MOSES)
Acronym: MOSES
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study did not get funded as anticipated
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2021-13414
Record Dates: First submitted 2023-02-17; First posted 2023-03-22 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Stroke (CVA) or TIA
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The study team will conduct a pragmatic comparative effectiveness study comparing standard stroke clinic follow up combined with RPM to aid with blood pressure management (n=30) versus standard stroke clinic follow, RPM and an added patient-facing smartphone application with educational modules and adherence incentives (n=30). Outcomes will include recruitment, retention and follow up metrics, self-reported adherence to medication regimens and life-style recommendations, patient engagement with RPM data and patient-facing application, cost-effectiveness of the interventions and changes in blood pressure as well as biomarkers such as HbA1c or LDL cholesterol levels. We hypothesize that RPM combined with a patient-facing application will improve patient reported and clinical outcomes of interest in the post-stroke transition of care setting.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): standard stroke clinic follow, combined with remote patient blood pressure monitoring and an added patient-facing smartphone application with educational modules and adherence incentives (n=30).
  Interventions: Behavioral: Standard of care, RPM and digital feedback
- Control arm (Active Comparator): standard stroke clinic follow up combined with remote blood pressure monitoring
  Interventions: Behavioral: Standard of care and RPM only

INTERVENTIONS:
Behavioral: Standard of care, RPM and digital feedback — Standard stroke follow up, RPM and a patient facing smartphone application containing real time BP feedback, educational models, treatment adherence push notification reminders, digital education and digital incentives (n=30). Outcomes will include recruitment, retention and follow up metrics, self-reported adherence to medication regimens and life-style recommendations, patient engagement with RPM data and patient-facing application, cost-effectiveness of the interventions and changes in blood pressure as well as biomarkers like LDL and Hemoglobin A1C.
  Arms: Intervention arm
Behavioral: Standard of care and RPM only — Standard stroke clinic follow up and remote blood pressure monitoring (n=30). Outcomes will include qualitative patient and provider experiences with the TBIs including barriers and facilitators to the use of RPM and patient-facing application in the study population
  Arms: Control arm

SUMMARY:
Despite decades of national declines in stroke incidence, racial/ethnic and socioeconomic disparities in stroke prevalence and care remain pervasive and the gap in these disparities is widening. Those who identify as African American (AA) or Hispanic are 2-3 times more likely to have a stroke when compared to those who identify as non-Hispanic White (NHW) and are also less likely to receive guideline-based medical therapy (e.g. mechanical thrombectomy, intravenous thrombolysis, discharge antithrombotic/anticoagulant, smoking cessation education) after their stroke. Additionally, people living in underserved communities with high local social deprivation indices and decreased community-level healthcare access, have an increased population-level risk of stroke. These inequities are likely multi-factorial and in large part related to decreased access to health promotion and preventive care services, as well as social/economic constraints impeding patients' access and compliance with medical treatment recommendations. Innovations in patient-facing digital health technologies, such as telemedicine, remote patient monitoring (RPM), and patient-facing smart phone applications could help bridge the gaps in post stroke care in marginalized communities by providing more accessible, convenient and perhaps effective, health care services. A recent secondary stroke prevention trial with predominantly African American and Hispanic participants compared blood pressure control measured by RPM combined with telehealth support vs. standard office-based follow up and found improved adherence and risk factor control in the digitally assisted group. However, there is limited knowledge around the patient and provider-level barriers, and supportive and educational resources needed to translating these and other similar findings into practice, especially in high-risk communities. Importantly, the same barriers to adopting digitally assisted care delivery during transitions of care and in the management of high-risk groups are shared across a number of episodic (e.g. ACS), acute on chronic (e.g. asthma, COPD, heart failure, DKA) and chronic diseases (e.g. hypertension, renal failure).

DETAILED DESCRIPTION:
Studying the implementation and uptake of technology based interventions (TBIs) after acute stroke hospitalization, may offer an ideal touch point to better understanding common translational bottlenecks to adopting TBIs across a number of other healthcare settings. Multiple Organized Systems for Engaging Stroke (MOSES) will employ a pragmatic comparative effectiveness design to study standard stroke clinic follow up combined with RPM for blood pressure management and compare it to standard clinic follow, RPM and an added patient-facing smartphone application with educational modules and adherence incentives. The investigator team hypothesizes that combining RPM with a patient-facing application consisting of treatment adherence reminders, digital education and digital incentives, will lead to improved care delivery and better compliance. Additionally, patient and user-centered outcomes, as well as perceived barriers to implementation by key stakeholders, will be studied. If successful, MOSES could improve the understanding of shared translational barriers related to implementation and uptake of TBIs in high-risk populations during transitions of care. Insights may also be applicable to the use of non blood pressure RPM, such as in digital scales, glucometers and sleep study devices. The investigator team plans to test this hypothesis and study patient-centered outcomes through the following two AIMS:

Specific Aims Aim1: To develop a culturally tailored patient facing application as an ancillary educational resource to using RPM and to aid with treatment plan adherence in the transition of care after acute stroke. In months 1-3, the study team plans to adapt a culturally tailored patient-facing smartphone application already being used in diabetes care (DiabetesXcel - developed by the research team at Montefiore-Einstein); to provide education on risk factor control strategies including use of RPM, treatment adherence push notification reminders, and digital incentives (gamification vs non-fungible tokens) in patients with recent hospitalization for acute stroke (secondary stroke prevention). Using a mixed methods approach feedback on the use of RPM and resources to be provided as part of a smart phone applications from 10 patients and 5 providers will be elicited, including potential unanticipated or undesirable effects. This patient and provider-centered analyses of TBIs (RPM, digitally delivered feedback regarding BP, digital incentives) will be performed in the Montefiore Comprehensive Stroke Center (CSC) clinic setting. Outcomes will include qualitative patient and provider experiences with the TBIs including barriers and facilitators to the use of RPM and patient-facing application in the study population. The investigator team hypothesizes that TBIs in the form of RPM and patient facing applications will be associated with a high level of patient and provider satisfaction.

Aim 2: To evaluate the impact of remote patient monitoring (RPM) and a patient-facing application on health outcomes in patients with recent TIA or minor stroke. In months 4-10, the investigator team will conduct a pragmatic comparative effectiveness study comparing standard stroke clinic follow up combined with RPM to aid with blood pressure management (n=30) versus standard stroke clinic follow, RPM and an added patient-facing smartphone application with educational modules and adherence incentives (n=30). Outcomes will include recruitment, retention and follow up metrics, self-reported adherence to medication regimens and life-style recommendations, patient engagement with RPM data and patient-facing application, cost-effectiveness of the interventions and changes in blood pressure as well as biomarkers such as HbA1c or LDL cholesterol levels. The study team hypothesizes that RPM combined with a patient-facing application will improve patient reported and clinical outcomes of interest in the post-stroke transition of care setting.

Approach Overall, the outcomes for each of the study aims will allow for a comprehensive understanding of the impact of RPM and a patient-facing application on health outcomes, as well as the barriers and facilitators to implementation and the feasibility and acceptability of the interventions in a high-risk inner-city community. The mixed methods framework and comparative effectiveness approach will allow for both a quantitative and qualitative understanding of the complexity of implementing the TBIs in this population. Specifically, the study team will conduct focus group sessions with 10 patients and 5 providers in the stroke clinic (NP, MDs, administrators) to gauge perceived digital health needs and value, as well as perceived barriers to TBI use. This values inventory-or the identification of where key beliefs and conceptions converge and diverge between these stakeholder groups is essential for avoiding unintended bias, unintended consequences, and can help advance the success of TBI interventions for preventative and chronic disease management. Further, the investigator team will conduct theory-informed formative and summative evaluation (e.g. perceived usefulness, ease of use) to aid in the understanding of the stakeholder's comfort and trust in various currently used and more novel TBIs including novel concepts and technologies which are increasingly influencing healthcare delivery (gamification, non-fungible tokens, smart contracts, machine learning, automation, decentralized autonomous organizations). The investigator team plans to use the information to improve functionality and usability of TBIs and to iteratively refine the RPM and patient facing application. To evaluate the process of TBI implementation in the Montefiore CSC clinic the study team will use the RE-AIM framework to assess the intervention's Reach (recruitment and retention rates, representativeness of the study sample),

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of recent TIA (<6 months) or minor stroke
* discharged to home with stroke clinic follow up planned
* modified Rankin score <3 at time of discharge.

Exclusion Criteria:

* Cognitive impairment limiting compliance with the intervention
* Modified Rankin score >2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
patient satisfaction | 1 month
  Telehealth Usability Questionnaire (TUQ) This is a 21 question survey which assesses 5 domains (usefulness, ease of use, reliability, effectiveness, satisfaction) of patient's satisfaction and usability of remote monitoring.
  Each question is ranked from 1-7 with 7 defined as "strong agreement/satisfaction" Min score is 21, max score is 147. The higher the score the greater the satisfaction/usability
provider satisfaction | 1 month
  Telehealth Usability Questionnaire (TUQ) This is a 21 question survey which assesses 5 domains (usefulness, ease of use, reliability, effectiveness, satisfaction) of a provider's satisfaction and usability of remote monitoring.
  Each question is ranked from 1-7 with 7 defined as "strong agreement/satisfaction" Min score is 21, max score is 147 The higher the score the greater the satisfaction/usability
compliance with medical follow up and treatment plan | 1 month
  defined by the number of telehealth visits over the course of the study Min is 0 and max is 10
medical knowledge of stroke symptoms | 1 month
  ability to identify the symptoms of stroke defined by the BEFAST Criteria. Min is 0, max is score 6, with higher score defined as having greater medical knowledge of stroke symptoms

SECONDARY OUTCOMES:
BP control | 1 month
  the weekly average systolic, diastolic blood pressure, and mean arterial pressure over the course of the study. All weekly measures will be averaged. Any erroneous values that fall 2 standard deviations away from the mean will be excluded.
  there is no min or max.
readmission rate | 30 days
  readmission rate for stroke or other acute illness at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Charles Esenwa, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: Undecided